CLINICAL TRIAL: NCT03332134
Title: Primary Prevention of Intimate Partner Violence in India
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National AIDS Research Institute, India (Unknown)
Responsible Party: Principal Investigator, Ameeta Kalokhe, Assistant Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00069846
Record Dates: First submitted 2017-11-02; First posted 2017-11-06 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Intimate Partner Violence
MeSH Terms: interventions — Poliovirus Vaccine, Inactivated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Married Couple Dyad (Experimental): Husband-wife dyads will receive the intimate partner violence (IPV) intervention program over the course of six weeks.
  Interventions: Behavioral: Intimate Partner Violence (IPV) Prevention Intervention
- Control Group (No Intervention): Husband-wife dyads in the control group will not receive an intervention.

INTERVENTIONS:
Behavioral: Intimate Partner Violence (IPV) Prevention Intervention — The IPV intervention consists of six sessions. Each session will cover one of 6 major modules to enhance transformation of motivation: 1) You, Me, and Us: Spending Meaningful Time Together, 2) I'm a Champion: I Can't Be Broken and I don't Accept Defeat! 3) Building Communication and conflict management strategies, and 4) Empowerment of the Couple: Planning Ahead, 5) Sexual communication and the sexual relationships, and 6) A Lens into Domestic Violence. The sessions will be audio-recorded and include a combination of didactics, interactive discussions, media use, and role play. The expected durations of session 1, 2-6, and the 3-month follow-up are 120 minutes, and 60-90 minutes, respectively.
  Arms: Married Couple Dyad

SUMMARY:
The goal of this study is to test and evaluate the feasibility, acceptance, safety, and efficacy of an an intimate partner violence (IPV) intervention in recently-married, low-income husband-wife dyads in Pune, India.

DETAILED DESCRIPTION:
The goal of this study is to test and evaluate the feasibility, acceptance, safety, and efficacy of an an intimate partner violence (IPV) intervention in recently-married, low-income husband-wife dyads in Pune, India conducted over a six week period.

Acceptability and feasibility will be assessed through semi-structured interviews with participants and staff post-intervention. Safety will be gauged through semi-structured interviews with women participants and efficacy will be gauged through change in proximal determinants of IPV in this population (i.e. time spent in the relationship, self-esteem, resilience, communication and conflict management skills, sexual communication, attitudes toward IPV acceptability, and conceptualization of IPV).

ELIGIBILITY:
Inclusion Criteria:

* Recently married (i.e. <1 year) husband-wife dyads
* First marriage
* Planning to reside in Pune for the majority of the next 6 months
* Marathi fluency
* Lives with partner
* Lives in a slum, slum redevelopment community, or chawl

Exclusion Criteria:

* Pregnant in third trimester of pregnancy
* Women who respond affirmatively to either a physical and/or sexual IPV item on the IFVCS short form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2018-10-09 (Actual); Study Completion 2018-10-09 (Actual)

PRIMARY OUTCOMES:
IPV Intervention Acceptability | Duration of Study (Up to 3 Months)
  Acceptability of the intervention to the dyad will be collected qualitatively and gauged by extracting themes regarding acceptability of modular content, timing of the intervention, safety precautions, number and duration of the intervention sessions, and appropriateness of intervention staff through semi-structured interviews between administrators and participants.
IPV Intervention Feasibility | Duration of Study (Up to 3 Months)
  Intervention feasibility will be qualitatively assessed by extracting themes from post-session semi-structured interviews of difficulties in intervention delivery, participant understanding of the intervention, and logistical problems with the intervention setting, timing, staff training, and debriefings as reported by the intervention administrator.
IPV Intervention Safety | Duration of Study (Up to 3 Months)
  Safety of the intervention will be gauged by extracting themes of incident IPV events or changes in IPV frequency or severity reported by the wife at the three-month follow-up through semi-structured interviews between administrators and participants.

SECONDARY OUTCOMES:
Change in Time Spent Together | Baseline, Post-Intervention (3 Months)
  Change in time spent together alone with partner
Change in Self-esteem | Baseline, Post-Intervention (3 Months)
  Change in score on Rosenberg Self-esteem Scale. The scale measures self-esteem on a scale of 0-30 (wherein lower scores are suggestive of lower self-esteem).
Change in Communication Skills | Baseline, Post-Intervention (3 Months)
  Change in confidence in communicating about various commonly-encountered scenarios with partner
Change in Conflict Negotiation Skills | Baseline, Post-Intervention (3 Months)
  Change in Revised Conflict Tactics Scale (CTS2) Negotiation Subscale score. The negotiation subscale measure actions taken to settle disagreements. The minimum score is 0 and the maximum is 150, with higher scores suggestive of better negotiation skills.
Change in Sexual Communication Skills | Baseline, Post-Intervention (3 Months)
  Change in confidence in communicating to partner desire to have or not have sex
Change in Reproductive Health Beliefs linked to IPV | Baseline, Post-Intervention (3 Months)
  Change in commonly held sexual and reproductive health beliefs linked to IPV perpetration.
Change in Conceptualization of IPV | Baseline, Post-Intervention (3 Months)
  Change in acknowledgement of behaviors that constitute IPV. This outcome is assessed using an adaptation of the Indian Family Violence and Control Scale, wherein response choices will include "not violence," "mild violence," "moderate violence, and "severe violence." The minimal score will be 12 and the maximum 48, with greater scores being suggestive of the participant having a more comprehensive conceptualization of behaviors constituting IPV.
Change in Attitudes toward IPV Acceptability | Baseline, Post-Intervention (3 Months)
  Change in attitudes toward situations in which beating a partner may be acceptable. This outcome is assessed using adapted questions from the National Family Health Survey Attitudes Towards Wife Beating module. It is assessed based on the frequency of affirmative responses to the questions, with more affirmative responses being associated with greater acceptance of IPV.

CONTACTS AND LOCATIONS:
Overall Officials: Ameeta Kalokhe, MD, Principal Investigator — Emory University
Locations (1):
- National AIDS Research Institute, Pune, Maharashtra, India

REFERENCES:
- [Derived] Kalokhe AS, Iyer S, Gadhe K, Katendra T, Kolhe A, Rahane G, Stephenson R, Sahay S. A Couples-Based Intervention (Ghya Bharari Ekatra) for the Primary Prevention of Intimate Partner Violence in India: Pilot Feasibility and Acceptability Study. JMIR Form Res. 2021 Feb 1;5(2):e26130. doi: 10.2196/26130. PMID 33459278
- [Derived] Kalokhe AS, Iyer S, Katendra T, Gadhe K, Kolhe AR, Paranjape A, Del Rio C, Stephenson R, Sahay S. Primary Prevention of Intimate Partner Violence Among Recently Married Dyads Residing in the Slums of Pune, India: Development and Rationale for a Dyadic Intervention. JMIR Res Protoc. 2019 Jan 18;8(1):e11533. doi: 10.2196/11533. PMID 30664483